CLINICAL TRIAL: NCT07287878
Title: Neural Mechanisms of Temporal Interference Stimulation on Improving Social Reward Function in Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22YF1439100
Record Dates: First submitted 2025-11-16; First posted 2025-12-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- orbitofrontal cortex (Experimental)
  Interventions: Device: Temporal Interference Simulation(TIS)
- parahippocampal gyrus (Experimental)
  Interventions: Device: Temporal Interference Simulation(TIS)
- striatum (Experimental)
  Interventions: Device: Temporal Interference Simulation(TIS)
- sham (Sham Comparator)
  Interventions: Device: Temporal Interference Stimulation(TIS)

INTERVENTIONS:
Device: Temporal Interference Simulation(TIS) — the total stimulation duration was 20 minutes, including a 40-second current ramp-up at the beginning and a 40-second ramp-down at the end.
  Arms: orbitofrontal cortex; parahippocampal gyrus; striatum
Device: Temporal Interference Stimulation(TIS) — Sham stimulation has only 40 seconds of current ramping-up and ramping-down at the beginning and end of the stimulation to simulate the sensation of actual stimulation.
  Arms: sham

SUMMARY:
Major depressive disorder (MDD) is a mood disorder characterized primarily by low mood, diminished interest, and reduced energy. Traditional views considered depression a non-degenerative condition; however, recent epidemiological studies have revealed its significant association with impaired social functioning. Data indicate that 59.3% of patients with depression experience social dysfunction of varying severity [1], particularly manifesting as difficulties in social interaction and relationship maintenance [2]. Therefore, investigating the mechanisms underlying social dysfunction is of great importance for promoting functional recovery in MDD, and dysfunction within the social reward system may represent a core factor, though the specific neural mechanisms remain unclear.

The ultimate goal of understanding the neural mechanisms underlying social reward impairment in depressed patients is to improve therapeutic outcomes. Temporal Interference (TI) stimulation, as a non-invasive deep brain stimulation technique, utilizes high-frequency current differentials to generate low-frequency amplitude-modulated electric fields, enabling precise targeting of deep brain regions. This study employs multimodal assessment methods-such as functional magnetic resonance imaging (fMRI), electroencephalography (EEG), and specific cognitive-behavioral tasks-combined with TI stimulation to observe immediate changes in functional connectivity, neural activity, and related cognitive functions (e.g., decision-making, memory) across participant groups. The research aims to elucidate the roles of the parahippocampal gyrus, orbitofrontal cortex, and striatum in social reward impairment in depression, and to explore circuit-based intervention targets, thereby providing novel strategies for the recovery of social functioning in MDD.

ELIGIBILITY:
Inclusion Criteria:

* 16-60 years old;
* Meeting with the criteria of major depressive disorder in the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5;
* Scored 20 or higher on the Hamilton's Depression Scale with 24 items (HAMD-24);
* With enough audio-visual ability and comprehensive ability to accomplish the visits;
* Be necessary and suitable to accept the treatment of antidepressants;
* Scored less than 14 on Hamilton's Anxiety Scale (HAMA) and scored less than 14 on the Hypomania Symptom Checklist-32 (HCL-32);
* With 2 or more atypical symptoms including significant weight gain or increase in appetite, hypersomnia, leaden paralysis, and a long-standing pattern of interpersonal rejection sensitivity that results in significant social or occupational impairment.

Exclusion Criteria:

* Severe medical or neurological problems;
* Previous mania or hypomania episodes;
* Female patients who are pregnant, planning to be pregnant or breastfeeding;
* Actively suicide ascertained by research psychiatrist or 3rd item of HAMD scored≥3(suicidality);
* Had ECT, MECT or rTMS in the past 6 months;
* Experienced severe personality disorder, mental retardation, anorexia/ bulimia nervosa.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HAMD) Score | baseline and immediately after the intervention
  The HAMD is a clinical depression assessment and consists of 17 items with a total score range from 0 to 54.A higher score indicates a worse outcome.
Change in The Positive and Negative Affect Schedule (PANAS) Score | Baseline and immediately after the intervention
  The Positive and Negative Affect Schedule (PANAS) is an assessment of participants' immediate affective states and consists of 20 items divided into two subscales (10 items for Positive Affect and 10 items for Negative Affect), with each item rated on a 5-point scale; higher scores on the Positive Affect subscale indicate more positive emotional states, while higher scores on the Negative Affect subscale indicate more negative emotional states.

SECONDARY OUTCOMES:
MRI measures | Baseline and immediately after the intervention
  The functional connectivity between stimulated target and the whole brain areas

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: Undecided